CLINICAL TRIAL: NCT01736696
Title: Phase 1, Investigator-Blind, Subject-Blind, Sponsor-Open, Placebo-Controlled, Two-Week, Multiple Dose Escalation Study In Medically Stable Subjects With Psoriasis To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of CP-690,550
Brief Title: Multiple Dose Escalation Study In Medically Stable Subjects With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921003
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis; Immunomodulation
Keywords: Psoriasis; PASI; plaques; skin biopsy; immunomodulation
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 5 mg BID (Experimental): 5 mg BID for 13 days and once on Day 14
  Interventions: Drug: tofacitinib
- 10 mg BID (Experimental): 10 mg BID for13 days and once on Day 14*
  Interventions: Drug: tofacitinib
- 20 mg BID (Experimental): 20 mg BID for 13 days and once on Day 14
  Interventions: Drug: tofacitinib
- 30 mg BID (Experimental): 30 mg BID for 13 days and once on Day 14
  Interventions: Drug: tofacitinib
- 60 mg QD (Experimental): 60 mg QD for 14 days
  Interventions: Drug: tofacitinib
- 50 mg BID (Experimental): 50 mg BID x 13 days and once on day 14
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — 5 mg BID For 13 days and once on Day 14
  Arms: 5 mg BID
Drug: tofacitinib — 10 mg BID for 13 days and once on Day 14*
  Arms: 10 mg BID
Drug: tofacitinib — 20 mg BID for 13 days and once on Day 14
  Arms: 20 mg BID
Drug: tofacitinib — 30 mg BID for 13 days and once on Day 14
  Arms: 30 mg BID
Drug: tofacitinib — 60 mg tablet once a day (QD) for 14 days
  Arms: 60 mg QD
Drug: tofacitinib — 50 mg tablets two times a day (BID) for 13 days and once on day 14
  Arms: 50 mg BID

SUMMARY:
This study was conducted in subjects with psoriasis to evaluate drug activity in this patient population by analysis of changes in psoriatic lesion biopsy characteristics. This subject population was selected to evaluate potentially relevant biological activity of CP-690,550 as well as assessing safety and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 18 and 65 years, inclusive, with active psoriasis lesion(s).
* Subjects should be healthy with the exception of psoriasis, where healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination. Blood pressure must be < 140/89. Body Mass Index (BMI) between 18-36 kg/m2, inclusive; and a total body weight >50 kg (110 lbs)
* The following laboratory variables must be no more than 10% below the lower limit of the normal reference range: RBC, hemoglobin, hematocrit, WBC, absolute neutrophil count. The absolute lymphocyte count must be greater than or equal to the lower limit of the reference range. Values for AST, ALT, bilirubin and alkaline phosphatase must be no more than 10% above the upper limit of the normal reference range. Values for total cholesterol and LDL must be no more than 20% above the upper limit of the normal reference range except for subjects being treated for hyperlipidemia. Normal glomerular filtration rate (> 80 mL/min).

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, urological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic disorder.
* Subjects with controlled essential hypertension and/or hyperlipidemia may be eligible for the study provided that any medications that are administered.
* Screening 12-lead ECG demonstrating at least one of the following: heart rate > 100 bpm, QRS >120 msec, QTc > 430 msec (males), QTc > 450 msec (females) or PR > 220 msec.
* Abnormal chest radiographs including, but not limited to, evidence of past or present tuberculosis infection. History of tuberculosis without treatment and/or positive tuberculin reaction without known vaccination with BCG.
* Subjects with a history of tumors with the exception of adequately treated basal cell carcinoma of the skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2002-11; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Little Rock, Arkansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921003&StudyName=Multiple%20Dose%20Escalation%20Study%20In%20Medically%20Stable%20Subjects%20With%20Psoriasis%20

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg (Cohort 1): CP-690,550 5 milligram (mg) oral powder for constitution (OPC) twice daily for 13 days and single oral dose on Day 14.
- CP-690,550 10 mg (Cohort 2): CP-690,550 10 mg OPC twice daily for 13 days and single oral dose on Day 14.
- CP-690,550 20 mg (Cohort 3): CP-690,550 20 mg OPC twice daily for 13 days and single oral dose on Day 14.
- CP-690,550 30 mg (Cohort 4): CP-690,550 30 mg OPC twice daily for 13 days and single oral dose on Day 14.
- CP-690,550 60 mg (Cohort 5): CP-690,550 60 mg tablets orally once daily up to Day 14.
- CP-690,550 50 mg (Cohort 6): CP-690,550 50 mg tablets orally twice daily for 13 days and single oral dose on Day 14.
- Placebo: Placebo matched to CP-690,550 for 13 days and single oral dose on Day 14.
Period: Overall Study
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Started | 5 | 5 | 10 | 9 | 9 | 8 | 13
Completed | 5 | 5 | 9 | 9 | 9 | 8 | 13
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13 | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.8) | 43.8 (7.4) | 39.6 (11.1) | 44.6 (11.1) | 46.9 (10.2) | 47.1 (9.7) | 44.4 (10.4) | 43.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 1 | 4 | 4 | 5 | 22
  Male | 2 | 3 | 7 | 8 | 5 | 4 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in QT Interval at 1 Hour Post Morning Dose (HPD 1) on Day 1
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2 minutes) were performed and average was calculated.QT interval: The time corresponding to the beginning of depolarization to repolarization of the ventricles. For each scheduled hour post morning dose (HPD), except for HPD=0, the time-matched baseline QT was defined as the mean of the triplicates on Day 0 at the same nominal HPD.
Time Frame: 23 hours (hrs) prior to morning dose on Day 1 (Baseline for HPD 1), 1 hour (hr) post morning dose on Day 1
Population: Analysis population included all participants who met the eligibility criteria.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
millisecond (msec)
  Baseline for HPD 1 | 372.20 (34.3) | 348.47 (23.52) | 369.40 (19.47) | 375.74 (24.65) | 383.96 (18.10) | 371.29 (28.33) | 370.95 (18.00)
  Change at HPD 1 on Day 1 | -6.33 (25.91) | 15.73 (9.04) | -6.33 (21.67) | 2.70 (14.54) | 1.63 (14.09) | -2.79 (13.28) | -4.21 (12.61)

2. Primary Outcome: Change From Baseline in QT Interval at 2 Hour Post Morning Dose (HPD 2) on Day 1
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated.QT interval: The time corresponding to the beginning of depolarization to repolarization of the ventricles. For each scheduled hour post morning dose (HPD), except for HPD=0, the time-matched baseline QT was defined as the mean of the triplicates on Day 0 at the same nominal HPD.
Time Frame: 22 hrs prior to morning dose on Day 1 (Baseline for HPD 2), 2 hrs post morning dose on Day 1
Population: Analysis population included all participants who met the eligibility criteria.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
msec
  Baseline for HPD 2 | 369.67 (33.78) | 350.27 (20.76) | 372.87 (21.10) | 377.48 (24.26) | 387.00 (18.81) | 374.00 (26.75) | 369.87 (17.53)
  Change at HPD 2 on Day 1 | -0.40 (26.39) | 9.80 (13.71) | -6.90 (22.22) | -0.15 (12.82) | -0.07 (9.40) | -1.58 (13.66) | -2.05 (16.76)

3. Primary Outcome: Change From Baseline in QT Interval at 4 Hour Post Morning Dose (HPD 4) on Day 1
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated.QT interval: The time corresponding to the beginning of depolarization to repolarization of the ventricles. For each scheduled HPD, except for HPD=0, the time-matched baseline QT was defined as the mean of the triplicates on Day 0 at the same nominal HPD.
Time Frame: 20 hrs prior to morning dose on Day 1 (Baseline for HPD 4), 4 hrs post morning dose on Day 1
Population: Analysis population included all participants who met the eligibility criteria. Here, the 'n' is signifying those participants who were evaluable for this measure at the specified time point for each arm group.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
msec
  Baseline for HPD 4 (n=5,5,10,9,9,8,13) | 373.73 (31.71) | 348.07 (23.34) | 373.20 (21.78) | 373.15 (20.46) | 381.44 (20.02) | 381.17 (26.96) | 368.00 (18.04)
  Change at HPD 4 on Day 1 (n=5,5,9,9,9,8,13) | -4.53 (23.17) | 11.53 (12.32) | 2.19 (20.98) | 2.96 (17.94) | 7.74 (14.69) | -8.17 (14.32) | -2.82 (10.82)

4. Primary Outcome: Change From Baseline in QT Interval at 8 Hour Post Morning Dose (HPD 8) on Day 1
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated.QT interval: The time corresponding to the beginning of depolarization to repolarization of the ventricles.For each scheduled HPD, except for HPD=0, the time-matched baseline QT was defined as the mean of the triplicates on Day 0 at the same nominal HPD.
Time Frame: 16 hrs prior to morning dose on Day 1 (Baseline for HPD 8), 8 hrs post morning dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
msec
  Baseline for HPD 8 (n=5,5,10,9,9,8,13) | 364.13 (36.00) | 356.73 (25.62) | 366.90 (22.02) | 374.56 (22.73) | 378.15 (23.91) | 372.25 (28.29) | 367.56 (17.95)
  Change at HPD 8 on Day 1 (n=5,5,9,9,9,8,13) | -1.27 (15.93) | -6.60 (10.71) | -3.96 (18.54) | -3.44 (12.75) | 7.67 (16.08) | -9.83 (15.12) | -9.03 (11.52)

5. Primary Outcome: Change From Baseline in QT Interval at 12 Hour Post Morning Dose (HPD 12) on Day 1
Description: as for outcome 4
Time Frame: 12 hrs prior to morning dose on Day 1 (Baseline for HPD 12), 12 hrs post morning dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
msec
  Baseline for HPD 12 (n=5,5,10,9,9,8,13) | 371.73 (31.50) | 351.27 (22.90) | 372.63 (22.54) | 370.11 (25.70) | 379.78 (24.93) | 363.08 (31.21) | 361.54 (16.29)
  Change at HPD 12 on Day 1 (n=5,5,9,9,9,8,13) | -6.27 (19.05) | -2.60 (5.27) | -4.15 (17.90) | 0.15 (9.79) | -3.22 (19.73) | -2.88 (14.01) | -1.36 (13.60)

6. Primary Outcome: Change From Baseline in QT Interval at 16 Hour Post Morning Dose (HPD 16) on Day 1
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated.QT interval: The time corresponding to the beginning of depolarization to repolarization of the ventricles.For each scheduled HPD, except for HPD=0, the time-matched baseline QT was defined as the mean of the triplicates on Day 0 at the same nominal HPD.Change from baseline in QT interval at HPD 16 was planned to be analyzed for participants who received CP-690,550 60 mg and matching placebo.
Time Frame: 8 hrs prior to morning dose on Day 1 (Baseline for HPD 16), 16 hrs post morning dose on Day 1
Population: Analysis population included all participants who met the eligibility criteria. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 60 mg (Cohort 5) | Placebo
Number analyzed (Participants) | 9 | 3
msec
  Baseline for HPD 16 | 377.15 (19.50) | 345.44 (18.77)
  Change at HPD 16 on Day 1 | 11.19 (19.98) | 13.11 (7.26)

7. Primary Outcome: Change From Baseline in QT Interval at 0 Hour Post Morning Dose (HPD 0) on Day 14
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated.QT interval: The time corresponding to the beginning of depolarization to repolarization of the ventricles. The mean of the triplicates at HPD=0 on Day 1 will be defined as the baseline for HPD=0.
Time Frame: Hour 0 (pre-dose) on Day 1 (Baseline for HPD 0), 0 hr on Day 14
Population: Analysis population included all participants who met the eligibility criteria.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
msec
  Baseline for HPD 0 | 374.80 (28.95) | 360.40 (28.03) | 367.70 (30.28) | 372.81 (27.83) | 383.41 (19.25) | 367.50 (22.12) | 364.03 (20.96)
  Change at HPD 0 on Day 14 | -14.53 (11.39) | 11.00 (12.00) | -0.33 (14.08) | 7.22 (16.38) | -9.70 (13.15) | -0.79 (17.48) | -7.08 (16.21)

8. Primary Outcome: Change From Baseline in QT Interval at 1 Hour Post Morning Dose (HPD 1) on Day 14
Description: as for outcome 4
Time Frame: 23 hrs prior to morning dose on Day 1 (Baseline for HPD 1), 1 hr post morning dose on Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
msec | -8.87 (12.12) | 22.27 (13.72) | 0.11 (12.55) | 2.81 (15.98) | -0.96 (14.63) | 0.71 (20.43) | -12.87 (17.82)

9. Primary Outcome: Change From Baseline in QT Interval at 2 Hour Post Morning Dose (HPD 2) on Day 14
Description: as for outcome 4
Time Frame: 22 hrs prior to morning dose on Day 1 (Baseline for HPD 2), 2 hrs post morning dose on Day 14
Population: Analysis population included all participants who met the eligibility criteria.'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
msec | -3.80 (12.18) | 18.67 (11.15) | -3.93 (13.21) | 6.89 (13.98) | -3.81 (17.18) | 2.46 (22.04) | -12.28 (19.35)

10. Primary Outcome: Change From Baseline in QT Interval at 4 Hour Post Morning Dose (HPD 4) on Day 14
Description: as for outcome 4
Time Frame: 20 hrs prior to morning dose on Day 1 (Baseline for HPD 4), 4 hrs post morning dose on Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
msec | -13.80 (15.37) | 6.53 (7.81) | -8.41 (7.25) | 18.96 (18.55) | 9.59 (10.70) | -4.79 (21.58) | -8.46 (21.09)

11. Primary Outcome: Change From Baseline in QT Interval at 8 Hour Post Morning Dose (HPD 8) on Day 14
Description: as for outcome 4
Time Frame: 16 hrs prior to morning dose on Day 1 (Baseline for HPD 8), 8 hrs post morning dose on Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
msec | -9.33 (11.31) | -0.53 (9.83) | -6.15 (15.86) | -1.96 (13.75) | 4.85 (18.51) | -2.67 (23.28) | -12.36 (11.38)

12. Primary Outcome: Change From Baseline in QT Interval at 12 Hour Post Morning Dose (HPD 12) on Day 14
Description: as for outcome 4
Time Frame: 12 hrs prior to morning dose on Day 1 (Baseline for HPD 12), 12 hrs post morning dose on Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
msec | -13.47 (12.76) | 8.00 (8.48) | -10.52 (10.63) | 0.81 (13.99) | -7.44 (22.73) | -0.63 (23.46) | -4.82 (15.31)

13. Primary Outcome: Number of Participants With Increase From Baseline in Corrected QT (QTc) Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum increase from baseline of 30 to less than (<) 60 msec(borderline) and greater than or equal to (>=) 60 msec (prolonged) were summarized.
Time Frame: 1, 2, 4, 8, 12 hrs post dose, additional 16 hrs post dose for 60 mg once daily group on Day 1; 1, 2 hrs post dose on Day 4, 7, 10;1,2,4,8,12 hrs post dose on Day 14; Day 21
Population: Analysis population included all participants who met the eligibility criteria.
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
participants
  QTcB,Maximum increase from baseline:30 to <60msec | 0 | 1 | 2 | 1 | 3 | 2 | 5
  QTcB,Maximum increase from baseline:>=60msec | 0 | 0 | 0 | 0 | 1 | 0 | 0
  QTcF,Maximum increase from baseline:30 to <60msec | 0 | 1 | 0 | 1 | 3 | 0 | 1
  QTcF,Maximum increase from baseline:>=60msec | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Corrected QT (QTc) Interval Greater Than or Equal to 500 Millisecond
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum QTc >=500 msec were reported.
Time Frame: as for outcome 13
Population: Analysis population included all participants who met the eligibility criteria.
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
participants
  QTcB | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) at Day 1
Description: AUCtau = area under the curve from time zero to end of dosing interval.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 1
Population: Pharmacokinetic analysis population included all participants who met the eligibility criteria and had 1 post-baseline pharmacokinetic assessment. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 9
nanogram*hour/milliliter (ng*hr/mL) | 161 (86.1) | 349 (34.7) | 732 (232) | 860 (235) | 2120 (837) | 1720 (453)

16. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) at Day 14
Description: AUCtau = area under the curve from time zero to end of dosing interval.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 4
ng*hr/mL | 154 (80.3) | 422 (49.5) | 850 (216) | 1350 (308) | 2600 (1580) | 1780 (501)

17. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) at Day 1
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 9
nanogram/milliliter (ng/mL) | 48.3 (24.5) | 90.5 (20.4) | 212 (62.3) | 180 (53.1) | 457 (88.2) | 429 (99.1)

18. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) at Day 14
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 4
ng/mL | 50.9 (21.2) | 87.7 (13.2) | 194 (53.9) | 225 (43.9) | 568 (205) | 403 (133)

19. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) at Day 1
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 1
Population: as for outcome 15
Measure: Median (Full Range); unit: hr
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 9
hr | 0.50 [0.25 to 1.00] | 0.50 [0.50 to 1.00] | 0.50 [0.25 to 2.00] | 0.50 [0.50 to 3.00] | 1.00 [0.50 to 3.00] | 1.00 [0.50 to 2.00]

20. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) at Day 14
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 14
Population: as for outcome 15
Measure: Median (Full Range); unit: hr
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 4
hr | 0.50 [0.50 to 0.50] | 1.00 [0.50 to 1.00] | 0.50 [0.25 to 2.00] | 1.00 [0.50 to 4.00] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 2.00]

21. Primary Outcome: Accumulation Ratio (R0)
Description: Accumulation ratio was calculated as, R0 = area under the curve from time zero to end of dosing interval (AUCtau) on Day 14 divided by area under the curve from time zero to end of dosing interval (AUCtau) on Day 1.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12 hrs post dose on Day 1 and Day 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6)
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 4
Ratio | 0.974 (0.181) | 1.22 (0.203) | 1.22 (0.389) | 1.62 (0.343) | 1.16 (0.270) | 1.14 (0.176)

22. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 1
Description: Absolute cell counts of cluster of differentiation 3 (CD3): T lymphocytes, cluster of differentiation 4 (CD4): Helper/Inducer T- Lymphocytes reactive with Major Histocompatability Complex-II (MHC-II), and cluster of differentiation 8 (CD8): Suppressor/Cytotoxic T-lymphocyte reactive with Major Histocompatability Complex-I (MHC-I), cluster of differentiation 16/56 (CD16/56): natural killer Cells, cluster of differentiation 19 (CD19): B-Lymphocytes determined using FACS.Baseline defined as mean of samples collected during screening, visit in which biopsy was taken, at Day 0 and at 0 hour Day 1.
Time Frame: Baseline, 1 hr post-dose on Day 1
Population: Analysis population included all participants who met the eligibility criteria.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
percent change
  Change at Day 1: CD3 | -14.39 (14.6) | 12.02 (18.2) | 1.17 (17.7) | 12.44 (17.4) | 8.38 (23.9) | 12.83 (14.0) | 0.52 (16.5)
  Change at Day 1: CD4 | -18.48 (19.4) | 8.65 (23.5) | -4.29 (15.2) | 5.99 (15.6) | -1.13 (19.9) | 8.54 (10.7) | 1.35 (18.3)
  Change at Day 1: CD8 | -7.58 (11.0) | 26.05 (25.1) | 8.90 (22.1) | 18.34 (21.4) | 13.90 (21.9) | 25.44 (14.6) | 0.42 (16.5)
  Change at Day 1: CD16/56 | 11.22 (27.0) | 79.99 (33.7) | 81.44 (62.7) | 74.07 (38.6) | 104.44 (85.8) | 103.74 (21.2) | -9.72 (18.3)
  Change at Day 1: CD19 | -27.11 (16.7) | -4.02 (30.9) | -10.30 (18.1) | -8.23 (10.4) | -6.22 (29.9) | -0.66 (9.0) | -6.46 (22.4)

23. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 2
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 2
Population: Analysis population included all participants who met the eligibility criteria. 'N' (number of participants analyzed)=participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 2: CD3 | 8.88 (24.0) | 34.74 (27.4) | 23.93 (31.1) | 46.07 (31.4) | 14.05 (24.4) | 52.43 (34.3) | -5.18 (17.4)
  Change at Day 2: CD4 | 8.58 (26.7) | 33.29 (25.4) | 26.73 (31.9) | 44.17 (33.9) | 18.85 (34.9) | 55.80 (35.5) | -6.85 (18.0)
  Change at Day 2: CD8 | 12.67 (19.3) | 32.68 (30.1) | 19.68 (29.3) | 43.04 (29.1) | 16.96 (25.1) | 50.97 (30.4) | -4.17 (20.2)
  Change at Day 2: CD16/56 | 18.27 (30.4) | 61.26 (47.8) | 52.84 (54.8) | 63.21 (45.1) | 0.61 (37.7) | 103.79 (45.8) | 5.61 (35.7)
  Change at Day 2: CD19 | 7.58 (40.3) | 9.56 (30.5) | 17.40 (24.5) | 30.39 (11.3) | 7.04 (33.5) | 45.72 (44.4) | -4.22 (24.4)

24. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 4
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 4
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 4: CD3 | -15.29 (21.1) | 51.71 (31.4) | 29.11 (49.0) | 71.55 (44.5) | 34.28 (41.8) | 32.81 (28.0) | 3.80 (28.2)
  Change at Day 4: CD4 | -15.87 (22.4) | 43.87 (22.0) | 30.90 (51.7) | 72.02 (43.1) | 42.50 (56.7) | 39.46 (27.2) | 6.08 (31.3)
  Change at Day 4: CD8 | -10.94 (17.8) | 56.72 (43.5) | 18.18 (41.7) | 61.61 (41.4) | 31.95 (32.6) | 29.81 (33.5) | -0.31 (24.8)
  Change at Day 4: CD16/56 | -23.08 (22.5) | 90.73 (41.6) | 10.67 (44.3) | 24.27 (55.5) | -5.23 (43.2) | -1.66 (44.8) | 7.18 (59.8)
  Change at Day 4: CD19 | -12.59 (27.2) | 41.44 (18.2) | 53.84 (71.8) | 56.27 (35.1) | 44.76 (55.7) | 77.25 (50.7) | -2.55 (37.5)

25. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 7
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 7
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 7: CD3 | 5.72 (20.6) | 28.15 (26.0) | 13.47 (55.4) | 25.51 (38.9) | 1.61 (26.0) | 34.77 (33.1) | -3.08 (17.3)
  Change at Day 7: CD4 | 6.52 (22.6) | 29.39 (22.2) | 14.99 (56.6) | 24.48 (39.3) | 0.91 (26.6) | 37.42 (33.1) | -3.28 (17.8)
  Change at Day 7: CD8 | 6.76 (18.5) | 31.50 (42.3) | 7.21 (50.1) | 21.74 (37.5) | 1.74 (25.2) | 30.95 (27.8) | -3.10 (19.8)
  Change at Day 7: CD16/56 | -10.57 (14.3) | 29.97 (56.6) | 17.02 (83.0) | -1.43 (40.0) | -2.37 (56.4) | -7.95 (30.2) | 2.26 (35.2)
  Change at Day 7: CD19 | 13.01 (36.3) | 34.47 (24.6) | 55.54 (83.2) | 72.86 (67.4) | 15.14 (46.0) | 98.64 (102.9) | -2.40 (22.3)

26. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 10
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 10
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 10: CD3 | 5.70 (18.9) | 8.76 (35.7) | 12.47 (49.1) | 36.76 (43.8) | 11.30 (50.0) | 12.61 (30.6) | -3.69 (27.9)
  Change at Day 10: CD4 | 6.86 (20.9) | 16.87 (34.0) | 14.50 (50.8) | 38.22 (43.0) | 14.61 (54.4) | 16.85 (32.4) | -4.52 (27.5)
  Change at Day 10: CD8 | 5.34 (20.9) | 4.13 (39.8) | 0.68 (35.4) | 28.77 (40.5) | 16.81 (62.4) | 7.87 (20.1) | -4.14 (30.6)
  Change at Day 10: CD16/56 | -16.73 (29.3) | -25.53 (41.4) | -16.22 (22.8) | -33.38 (27.2) | -21.99 (36.1) | -37.90 (24.8) | -10.82 (31.3)
  Change at Day 10: CD19 | 24.06 (26.9) | 34.97 (38.7) | 76.05 (71.1) | 79.94 (69.2) | 63.64 (180.0) | 84.57 (109.7) | -13.19 (31.5)

27. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 14
Description: as for outcome 22
Time Frame: Baseline; hr 0, 8 hr post-dose on Day 14
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at 0 hr post dose on Day 14: CD3 | 1.01 (16.0) | 26.93 (21.5) | 7.07 (33.0) | 14.91 (32.1) | 10.74 (37.1) | 12.69 (43.9) | -15.05 (21.7)
  Change at 8 hr post dose on Day 14: CD3 | 7.98 (18.2) | 76.59 (28.7) | 19.79 (23.1) | 40.85 (36.7) | 44.08 (61.6) | 15.64 (32.3) | -7.20 (20.7)
  Change at 0 hr post dose on Day 14: CD4 | -1.91 (19.0) | 31.80 (11.0) | 9.86 (41.2) | 14.80 (32.3) | 9.67 (49.1) | 17.69 (46.8) | -15.51 (25.1)
  Change at 8 hr post dose on Day 14: CD4 | 7.31 (18.0) | 86.33 (30.3) | 22.68 (24.8) | 38.65 (36.7) | 57.94 (91.5) | 19.21 (30.4) | -5.88 (23.1)
  Change at 0 hr post dose on Day 14: CD8 | 6.92 (9.1) | 25.57 (37.0) | -3.36 (23.6) | 10.68 (30.9) | 17.58 (42.4) | 9.89 (35.5) | -14.21 (20.2)
  Change at 8 hr post dose on Day 14: CD8 | 10.36 (17.3) | 70.26 (34.0) | 16.37 (16.9) | 40.38 (34.4) | 42.59 (59.2) | 31.87 (86.9) | -6.94 (18.9)
  Change at 0 hr post dose on Day 14: CD16/56 | -0.34 (25.0) | 1.73 (52.8) | -28.06 (32.3) | -43.06 (21.4) | -20.03 (44.6) | -42.70 (35.0) | -6.49 (25.4)
  Change at 8 hr post dose on Day 14: CD16/56 | -8.06 (19.7) | 41.85 (47.4) | -6.44 (38.0) | -8.75 (46.5) | 45.94 (114.4) | -14.38 (37.9) | -4.09 (34.0)
  Change at 0 hr post dose on Day 14: CD19 | 16.76 (25.1) | 39.97 (33.3) | 69.43 (75.9) | 68.14 (72.2) | 60.99 (151.4) | 116.93 (215.8) | -16.04 (33.1)
  Change at 8 hr post dose on Day 14: CD19 | 20.74 (19.8) | 92.47 (47.9) | 117.56 (52.4) | 95.87 (86.6) | 78.60 (94.0) | 152.66 (263.6) | 2.53 (36.2)

28. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 18
Description: as for outcome 22
Time Frame: Baseline, Hour 0 on Day 18
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 8 | 8 | 13
percent change
  Change at Day 18: CD3 | 13.89 (27.9) | -14.04 (30.6) | -10.24 (21.3) | -10.65 (18.5) | -14.54 (13.5) | -46.69 (17.5) | 3.91 (20.0)
  Change at Day 18: CD4 | 12.44 (29.6) | -13.35 (24.9) | -7.80 (21.5) | -8.89 (17.4) | -13.66 (19.1) | -42.60 (18.8) | 7.17 (17.1)
  Change at Day 18: CD8 | 17.52 (32.7) | -9.18 (44.1) | -12.38 (23.1) | -18.76 (24.0) | -13.47 (8.0) | -51.68 (18.1) | 4.70 (15.9)
  Change at Day 18: CD16/56 | 11.58 (31.5) | -7.64 (73.7) | -21.03 (46.0) | -48.63 (63.5) | -17.13 (45.7) | -76.21 (28.2) | -0.68 (22.4)
  Change at Day 18: CD19 | 16.98 (50.8) | -15.78 (15.9) | 13.95 (32.5) | 22.65 (45.8) | -8.14 (35.6) | -29.44 (25.4) | -4.67 (25.8)

29. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 21
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 21: CD3 | -25.48 (10.5) | -6.38 (14.8) | -42.27 (23.9) | -14.82 (20.2) | -7.93 (13.5) | -27.37 (13.3) | -1.12 (17.8)
  Change at Day 21: CD4 | -29.75 (9.6) | -2.88 (7.4) | -41.01 (24.4) | -11.01 (20.7) | -9.41 (16.5) | -22.38 (13.1) | 1.16 (19.8)
  Change at Day 21: CD8 | -19.51 (14.0) | -6.00 (31.1) | -43.55 (28.9) | -23.78 (21.1) | -2.12 (14.8) | -32.49 (15.6) | -4.01 (17.8)
  Change at Day 21: CD16/56 | -7.23 (23.5) | -9.21 (63.8) | -47.87 (30.7) | -48.04 (19.0) | 5.62 (35.4) | -66.94 (19.2) | -2.22 (44.1)
  Change at Day 21: CD19 | -20.90 (25.4) | -14.61 (26.7) | -22.60 (26.6) | -7.67 (34.8) | -17.50 (27.7) | -12.51 (22.9) | 0.98 (24.3)

30. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 28
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 28
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 28: CD3 | -18.11 (10.0) | 9.29 (24.5) | 0.38 (34.1) | -4.60 (17.9) | -7.60 (23.3) | -22.08 (9.7) | -2.57 (25.0)
  Change at Day 28: CD4 | -21.29 (13.3) | 10.97 (29.8) | 1.02 (35.2) | -5.90 (15.7) | -11.51 (19.8) | -19.90 (6.3) | -2.86 (24.9)
  Change at Day 28: CD8 | -11.96 (9.0) | 11.58 (18.8) | -2.84 (35.0) | -9.33 (18.5) | -6.13 (21.8) | -23.56 (13.7) | -1.56 (26.7)
  Change at Day 28: CD16/56 | 5.13 (35.9) | 21.93 (51.3) | -10.27 (31.2) | -28.52 (51.6) | 11.21 (55.9) | -26.96 (39.4) | 13.32 (50.8)
  Change at Day 28: CD19 | -7.96 (24.3) | 21.29 (23.5) | 1.96 (42.3) | -6.53 (21.8) | -16.50 (28.3) | -11.58 (22.1) | -12.51 (19.1)

31. Primary Outcome: Percent Change From Baseline in Fluorescence-Activated Cell Sorting (FACS) Analysis at Day 42
Description: as for outcome 22
Time Frame: Baseline, hr 0 on Day 42
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
percent change
  Change at Day 42: CD3 | -20.79 (29.0) | -15.72 (29.9) | -11.58 (30.0) | -1.60 (19.5) | -9.17 (21.5) | -1.63 (20.2) | 0.19 (32.6)
  Change at Day 42: CD4 | -25.65 (30.3) | -19.27 (29.2) | -11.42 (30.0) | -4.08 (17.5) | -12.27 (24.6) | -3.81 (12.0) | 0.96 (35.7)
  Change at Day 42: CD8 | -12.74 (29.1) | -10.04 (37.2) | -12.93 (33.9) | -5.60 (19.8) | -3.24 (17.6) | 4.19 (31.4) | 3.57 (33.5)
  Change at Day 42: CD16/56 | -9.01 (25.4) | 21.15 (70.8) | -2.32 (27.9) | 2.87 (76.1) | 24.08 (35.8) | -4.54 (37.4) | 19.90 (41.5)
  Change at Day 42: CD19 | -31.86 (30.9) | 6.43 (33.6) | -9.39 (29.2) | -10.22 (27.3) | -20.20 (30.0) | -8.30 (16.8) | -3.93 (52.5)

32. Primary Outcome: Change From Baseline in Immune Cell Function at Day 14
Description: The degree of immunosuppression induced by the study drug administration was evaluated using a bioluminescent assay in which the concentration of Adenosine-5-Triphosphate (ATP) released by CD4 cells was measured. ATP concentrations released from stimulated and unstimulated cells were evaluated. ATP Concentration less than or equal to (<=) 225: low immune cell response, 226 to 524: Moderate immune cell response, >= 525: strong immune cell response. Baseline was defined as the mean of the samples collected during the pre-dose biopsy.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 14
Population: Analysis population included all participants who met the eligibility criteria. 'N' (number of participants analyzed)=participants evaluable for this measure. 'n' = participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 2 | 5 | 10 | 9 | 9 | 7 | 13
ng/mL
  Baseline: Stimulated ATP(n=2,5,10,9,9,7,13) | 222.75 (157.3) | 205.40 (143.1) | 429.00 (115.3) | 406.11 (171.6) | 210.56 (104.1) | 252.50 (146.3) | 301.88 (152.9)
  Baseline: Unstimulated(Uns) ATP(n=2,5,10,9,9,7,13) | 11.50 (9.9) | 10.60 (3.2) | 16.30 (6.6) | 16.44 (10.2) | 14.11 (8.3) | 7.14 (5.9) | 16.00 (12.4)
  Change at Day 14: Stimulated ATP(n=2,5,9,9,9,7,13) | 92.75 (120.6) | 95.80 (135.0) | 155.11 (168.0) | 90.11 (125.9) | 118.78 (88.2) | 61.21 (124.7) | 26.81 (66.6)
  Change at Day 14:Uns ATP(n=2,5,9,9,9,7,13) | 9.50 (2.8) | 5.60 (11.4) | 0.44 (8.9) | 0.33 (10.6) | 1.67 (15.4) | 0.29 (13.1) | 1.46 (11.2)

33. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 2
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 2
Population: Analysis population included all participants who met the eligibility criteria. 'n' = participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: 1000 cells/cubic millimeter (cells/mm^3)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 10 | 9 | 9 | 8 | 13
1000 cells/cubic millimeter (cells/mm^3)
  Baseline (n=5,5,10,9,9,8,13) | 124.00 (30.6) | 94.00 (36.9) | 81.50 (20.1) | 95.22 (14.3) | 80.56 (24.4) | 79.75 (25.8) | 100.69 (46.2)
  Change at Day 2 (n=5,5,9,9,8,8,12) | -6.60 (21.3) | -2.00 (13.7) | 20.00 (16.1) | -17.67 (24.2) | -10.88 (19.7) | -3.75 (11.1) | -7.25 (28.8)

34. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 4
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
1000 cells/mm^3 | -14.00 (17.2) | -7.60 (16.5) | 17.33 (26.6) | -48.44 (13.3) | -14.67 (16.4) | -20.00 (14.9) | -20.85 (41.2)

35. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 7
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
1000 cells/mm^3 | -3.40 (18.7) | 6.40 (15.9) | 17.11 (26.5) | -14.44 (13.6) | 3.22 (20.6) | -30.38 (13.8) | -1.38 (31.1)

36. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 10
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 12
1000 cells/mm^3 | -16.40 (29.5) | -14.00 (18.3) | 16.00 (25.9) | -18.22 (15.9) | 6.56 (17.5) | -29.50 (21.5) | -3.42 (38.8)

37. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 15
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 7 | 12
1000 cells/mm^3 | -24.00 (25.3) | -11.40 (17.4) | -8.56 (11.9) | -42.22 (16.9) | 24.11 (16.8) | -31.57 (25.9) | -17.92 (28.4)

38. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 21
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 6 | 13
1000 cells/mm^3 | -13.40 (30.6) | 17.60 (11.5) | 44.22 (27.1) | 5.44 (14.4) | 40.25 (15.6) | -9.17 (23.9) | 12.54 (40.2)

39. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 28
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 8 | 8 | 13
1000 cells/mm^3 | -16.20 (8.2) | 47.60 (14.8) | 49.56 (24.0) | 23.89 (23.5) | 21.75 (13.6) | 56.00 (24.1) | -2.85 (32.5)

40. Primary Outcome: Change From Baseline in Reticulocyte Count at Day 42
Description: Reticulocyte count was assessed to detect potential of Janus kinase 2 (JAK2) mediated erythropoiesis.
Time Frame: Baseline (Within 7 days prior to Day 1), Day 42
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
1000 cells/mm^3 | -4.60 (12.6) | -7.00 (35.9) | 34.56 (30.0) | -3.67 (12.5) | -2.33 (21.9) | 22.50 (31.7) | -18.00 (26.7)

41. Primary Outcome: Time to Reach Maximum Change From Baseline and Time to Return to Baseline Value for Fluorescence-Activated Cell Sorting (FACS), Reticulocyte Counts and Immune Cell Function
Time Frame: Day 0 (pre-dose), 1, 2, 4, 7, 10, 14, 15, 18, 21, 28, 42
Population: Data was not analyzed as per planned analyses due to pattern of changes observed.
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

42. Primary Outcome: Half Maximal Effective Area Under the Concentration-Time Curve 50 (EAUC 50)
Description: EAUC 50 was calculated from a regression analyses using area under the concentration-time curve (AUC) as the independent variable. A sigmoid maximum effect (Emax) model was used to explain the relationship between AUC and modified Psoriasis Severity Index (mPASI) score, where Emax was the maximum effect (100 percent reduction in the total mPASI score from baseline), and EAUC 50 was the AUC where 50 percent of the maximum effect was measured.
Time Frame: Day 14
Population: as for outcome 6
Measure: Number; unit: ng*hr/mL
Groups:
- All CP-690,550 Treated Participants: Included all participants who received either CP-690,550 OPC or CP-690,550 tablets for 14 days.
Arm/Group | All CP-690,550 Treated Participants
Number analyzed (Participants) | 45
ng*hr/mL | 2696

43. Secondary Outcome: Number of Participants With Modified Psoriasis Severity Index (mPASI) at Day 14
Description: Modified Psoriasis Area and Severity Index (mPASI) assessed lesion severity but not the body surface area affected. Severity was estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final mPASI = sum of the each component scores. Total score range 0-12 , higher score indicated more severity.
Time Frame: Baseline (Within 7 days prior to Day 1) up to Day 14
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
participants
  Erythema: 0 | 1 | 0 | 0 | 2 | 2 | 4 | 0
  Erythema: 1 | 3 | 4 | 8 | 7 | 4 | 4 | 4
  Erythema: 2 | 1 | 1 | 1 | 0 | 3 | 0 | 9
  Erythema: 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration: 0 | 0 | 1 | 3 | 4 | 1 | 6 | 1
  Induration: 1 | 2 | 3 | 5 | 3 | 6 | 0 | 2
  Induration: 2 | 2 | 1 | 1 | 2 | 2 | 2 | 9
  Induration: 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Induration: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Scaling: 0 | 0 | 1 | 1 | 0 | 2 | 5 | 0
  Scaling: 1 | 3 | 2 | 6 | 7 | 3 | 2 | 8
  Scaling: 2 | 2 | 2 | 2 | 2 | 4 | 1 | 4
  Scaling: 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Scaling: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With Physician's Global Assessment (PGA) of Psoriasis
Description: Physician global assessment (PGA) of Psoriasis is a 7-point scale used to assess severity of psoriatic plaques, scaling and/or erythema. Severity scale ranged from 1 to 7: 1=severe, 2=moderate to severe, 3=moderate, 4=mild to moderate, 5=mild, 6=almost clear, 7=clear (no sign of psoriasis).
Time Frame: Baseline (Within 7 days prior to Day 1) up to Day 14
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 9 | 9 | 9 | 8 | 13
participants
  PGA:1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PGA:2 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  PGA:3 | 3 | 1 | 3 | 2 | 0 | 0 | 5
  PGA:4 | 0 | 3 | 2 | 1 | 4 | 2 | 2
  PGA:5 | 1 | 0 | 2 | 4 | 3 | 0 | 5
  PGA:6 | 0 | 1 | 2 | 2 | 0 | 4 | 1
  PGA:7 | 0 | 0 | 0 | 0 | 1 | 2 | 0

45. Secondary Outcome: Gene Expression in Psoriatic Plaque Biopsies
Description: Gene expression by quantitative polymerized chain reaction (PCR) using standard curve (SC) method generated by linear regression using log threshold cycle versus log(cell number). Keratin (K)-16, inducible nitric oxide synthase (iNOS), Interleukin 8 (IL-8), CD25, Granzyme B, IL-2, IL-7, IL-15, Interferon-gamma (INF-gamma), C-X-C motif chemokine(CXCL10), perforin 1, B-cell Lymphoma 2 (BCL-2), BCL2 associated X Protein (BAX), Tumor Necrosis Factor Fas Ligand (TNF-FasL), and proliferating cell nuclear antigen (PCNA) presented as control gene normalized expression (relative expression) within SC.
Time Frame: Day 14
Population: Analysis population:all participants who met eligibility criteria. 'N'(number of participants analyzed)=participants evaluable for this measure. 'n =participants evaluable for specified category for each arm group respectively. Gene expression results were planned to be analyzed for participants who received CP-690,550 5,30 mg and matching placebo.
Measure: Mean (Standard Deviation); unit: relative expression unit (REU)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 30 mg (Cohort 4) | Placebo
Number analyzed (Participants) | 2 | 2 | 1
relative expression unit (REU)
  BCL-2 | 0.47 (0.09) | 0.36 (0.14) | 2.29 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  BAX | 1.16 (0.21) | 0.83 (0.28) | 0.68 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  CD25 | 7.34 (2.33) | 1.05 (0.27) | 0.16 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  CXCL10 | 15.03 (5.75) | 0.44 (0.45) | 0.04 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Granzyme B | 42.71 (18.54) | 1.20 (0.07) | 0.03 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  IL-2 | 0.98 (0.16) | 0.87 (0.02) | 0.75 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  IL-8 | 556.12 (754.91) | 14.66 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  INOS | 77.79 (40.10) | 0.97 (0.08) | 0.02 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  INF-gamma | 2.26 (1.49) | 0.90 (0.09) | 0.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  IL-15 | 0.51 (0.01) | 0.70 (0.06) | 0.86 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  IL-7 | 0.85 (0.11) | 1.26 (0.51) | 1.19 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  K-16 | 69.04 (7.60) | 5.18 (2.63) | 0.04 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  PCNA | 2.09 (0.77) | 1.15 (0.06) | 0.41 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Perforin | 2.80 (2.56) | 0.65 (0.17) | 0.23 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  TNF-FasL | 0.95 (0.24) | 1.24 (0.86) | 0.64 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

46. Secondary Outcome: Immunohistochemistry From Psoriatic Plaque Biopsies
Description: Immunohistochemical staining of skin biopsies was performed with monoclonal antibodies directed against cluster of differentiation 3 (CD3) and cluster of differentiation 8 (CD8) T-lymphocytes, cluster of differentiation 16/56 (CD16/56) natural killer cells, and cluster of differentiation 83 (CD83) mature dendritic cells. Baseline was defined as mean of samples obtained at the screening visit within 7 days prior to Day 1, at the baseline biopsy, and Day 0. Immunohistochemistry results were planned to be analyzed for participants who received CP-690,550 5, 20, 30 mg and matching placebo.
Time Frame: Baseline (within 7 days prior to Day 1), Day 14
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: cells/microliter (cells/μL)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | Placebo
Number analyzed (Participants) | 1 | 1 | 4 | 2
cells/microliter (cells/μL)
  Baseline: CD3 epidermal (n=1,1,4,2) | 115.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 108.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 122.50 (50.8) | 124.50 (55.9)
  Baseline: CD3 dermal (n=1,1,4,2) | 189.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 135.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 130.00 (81.3) | 196.00 (99.0)
  Baseline: CD8 epidermal (n=1,1,4,2) | 66.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 55.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 108.50 (40.9) | 71.50 (19.1)
  Baseline: CD8 dermal (n=1,1,4,2) | 23.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 53.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 123.75 (103.6) | 74.00 (70.7)
  Baseline: CD83 epidermal (n=1,1,4,2) | 13.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 44.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 17.00 (12.1) | 1.50 (0.7)
  Baseline: CD83 dermal (n=1,1,4,2) | 11.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 78.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 18.00 (7.3) | 3.00 (0.0)
  Baseline: Absolute CD16/56 (n=0,0,0,0) | NA (NA) — Data was not analyzed as per planned analyses. | NA (NA) — Data was not analyzed as per planned analyses. | NA (NA) — Data was not analyzed as per planned analyses. | NA (NA) — Data was not analyzed as per planned analyses.
  Day 14: CD3 epidermal (n=1,1,4,2) | 148.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 96.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 82.25 (121.0) | 97.00 (41.0)
  Day 14: CD3 dermal (n=1,1,4,2) | 120.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 114.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 95.25 (59.4) | 92.00 (53.7)
  Day 14: CD8 epidermal (n=1,1,4,2) | 85.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 56.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 51.50 (50.8) | 41.50 (34.6)
  Day 14: CD8 dermal (n=1,1,4,2) | 27.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 42.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 90.50 (54.4) | 25.00 (9.9)
  Day 14: CD83 epidermal (n=1,1,4,2) | 42.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.25 (1.5) | 7.00 (9.9)
  Day 14: CD83 dermal (n=1,1,4,2) | 26.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 17.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 3.25 (2.2) | 9.50 (9.2)
  Day 14: Absolute CD16/56 (n=0,0,0,0) | NA (NA) — Data was not analyzed as per planned analyses. | NA (NA) — Data was not analyzed as per planned analyses. | NA (NA) — Data was not analyzed as per planned analyses. | NA (NA) — Data was not analyzed as per planned analyses.

47. Secondary Outcome: Number of Participants With Keratin 16 (K16) Expression
Description: Immunohistochemical staining of skin biopsies was performed with monoclonal antibodies directed against K16. Number of participants with K16 expression were assessed qualitatively using suprabasal keratinocytes.
Time Frame: Baseline (within 7 days prior to Day 1) up to Day 14
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | Placebo
Number analyzed (Participants) | 1 | 1 | 4 | 2
participants
  Baseline | 1 | 1 | 4 | 2
  Day 14 | 1 | 1 | 4 | 2

48. Secondary Outcome: Number of Participants With Intracellular Adhesion Molecule (ICAM-1) by Epidermal Keratinocytes Expression
Description: Immunohistochemical staining of skin biopsies was performed with monoclonal antibodies directed against ICAM-1. Number of participants with ICAM-1 expression was to be assessed qualitatively using epidermal keratinocytes.
Time Frame: Baseline (within 7 days prior to Day 1) up to Day 14
Population: Analysis of ICAM-1 in biopsy specimens was not performed as it often continues to be expressed on vessels in the skin even when psoriasis was resolved, thus would not provide a measure of response to therapy.
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

49. Secondary Outcome: Gene Expression in Peripheral Blood
Description: Punch biopsy and serum blood were assayed for messenger Ribonucleic acid (mRNA) gene expression by quantitative PCR using standard curve(SC) method generated by linear regression using log threshold cycle versus log(cell number). granzyme B, IFN-gamma, TNF-alpha (FasL and superfamily member 5 [SF5]), BCL2, BAX, iNOS, and CD 25 presented as control gene normalized expression(relative expression) within SC. The Relative mRNA Gene Expression Level is relative to baseline and normalized to the housekeeping gene 18 Svedberg unit ribosomal RNA (18S rRNA).
Time Frame: Day 14
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: relative expression unit (REU)
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 30 mg (Cohort 4) | Placebo
Number analyzed (Participants) | 9 | 9 | 6
relative expression unit (REU)
  Granzyme B (n=9,9,6) | 0.69 (0.33) | 0.99 (0.58) | 1.58 (1.13)
  IFN-gamma (n=9,9,6) | 2.06 (1.58) | 1.16 (0.59) | 1.46 (0.86)
  TNF-SF5 (n=9,9,6) | 1.79 (1.14) | 1.29 (0.48) | 1.24 (0.38)
  TNF-FasL (n=9,9,6) | 0.99 (0.37) | 1.09 (0.53) | 1.27 (0.83)
  BCL2 (n=9,9,6) | 0.71 (0.40) | 0.90 (0.30) | 1.01 (0.22)
  BAX (n=9,9,6) | 1.10 (0.32) | 0.98 (0.25) | 0.97 (0.22)
  iNOS (n=2,1,1) | 77.79 (40.10) | 0.97 (0.08) | 0.02 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  CD 25 (n=9,9,6) | 1.19 (0.50) | 1.02 (0.29) | 1.01 (0.24)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 5 mg (Cohort 1) | CP-690,550 10 mg (Cohort 2) | CP-690,550 20 mg (Cohort 3) | CP-690,550 30 mg (Cohort 4) | CP-690,550 60 mg (Cohort 5) | CP-690,550 50 mg (Cohort 6) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/10 | 0/9 | 0/9 | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 3/10 | 1/9 | 2/9 | 2/8 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Cohort 1) (N=5) | CP-690,550 10 mg (Cohort 2) (N=5) | CP-690,550 20 mg (Cohort 3) (N=10) | CP-690,550 30 mg (Cohort 4) (N=9) | CP-690,550 60 mg (Cohort 5) (N=9) | CP-690,550 50 mg (Cohort 6) (N=8) | Placebo (N=13)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Cohort 1) (N=5) | CP-690,550 10 mg (Cohort 2) (N=5) | CP-690,550 20 mg (Cohort 3) (N=10) | CP-690,550 30 mg (Cohort 4) (N=9) | CP-690,550 60 mg (Cohort 5) (N=9) | CP-690,550 50 mg (Cohort 6) (N=8) | Placebo (N=13)
Headache (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2
Lab test abnormal (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Peripheral edema (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SGOT increased (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SGPT increased (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.